CLINICAL TRIAL: NCT07357298
Title: Phase III Trial of Brain MRI Surveillance in Stage IV Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Department of Health (Other Government); Florida Biomedical Research Program - Bankhead Coley (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MCC-24030
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surveillance Brain MRI (Other): Participants receive a baseline brain MRI followed by surveillance brain MRI every 6 months for 24 months.
  Interventions: Diagnostic Test: Surveillance Brain MRI
- Standard of Care Brain Imaging (Other): Participants receive a baseline brain MRI followed by standard-of-care imaging only if neurologic symptoms develop.
  Interventions: Diagnostic Test: Standard of Care Brain Imaging

INTERVENTIONS:
Diagnostic Test: Surveillance Brain MRI — Routine scheduled MRI imaging at baseline and at 6-month intervals.
  Arms: Surveillance Brain MRI
Diagnostic Test: Standard of Care Brain Imaging — Imaging performed only when clinically indicated.
  Arms: Standard of Care Brain Imaging

SUMMARY:
This randomized, multi-institutional phase III trial evaluates whether routine surveillance brain MRI every 6 months improves detection and treatment characteristics of brain metastases in neurologically asymptomatic patients with stage IV breast cancer. Patients are stratified by receptor subtype, age, prior therapy, and study site, then randomized 1:1 to either scheduled surveillance MRIs or standard-of-care symptom-triggered imaging. The study aims to determine whether earlier detection leads to differences in treatment modality, frequency of brain metastases, leptomeningeal disease incidence, quality of life, and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of breast cancer with documentation of ER/PR/HER2 status
* Radiographic evidence of stage IV extracranial disease enrolled within 60 days of diagnosis or starting first line therapy. HR+/HER2- patients may be enrolled within 60 days of starting 2nd line therapy as well.
* HR+ will be defined as ER and/or PR > 10%. To be classified as HER2+ disease, overexpression of HER2 by either IHC or in-situ hybridization is necessary as defined by the ASCO / CAP Guidelines41. Triple negative will be classified as ER and PR <10% and HER2-.
* Age ≥ 18
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group performance status ≤ 2
* Patients must be able to understand and the willingness to sign an informed consent for study procedures
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Prior diagnosis or treatment of brain metastases or leptomeningeal disease
* History of other non-breast malignancy requiring treatment with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as but not limited to, non-melanoma skin cancers, stage I endometrioid uterine cancer, and others at the discretion of the PI
* Neurologic symptoms warranting standard screening brain MRI in the judgement of the treating physician at time of enrollment
* Indications warranting brain MRI for other neurologic conditions at time of study entry (including multiple sclerosis, stroke, traumatic brain injuries, epilepsy, hydrocephalus and pituitary gland disorders)
* Contraindication towards MRI with contrast
* Chronic kidney disease stage IV or V or end stage renal disease (CrCl <30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Treatment Characteristics of Brain Metastases | Up to 24 Months
  Proportion of patients receiving surgery or whole-brain radiation therapy for brain metastases.

SECONDARY OUTCOMES:
Frequency of Brain Metastases | Up to 24 Months
  The frequency of metastasis detection over the 24-month screening/follow-up period.
Leptomeningeal Disease Incidence | Up to 24 Months
  Incidence of radiographic detection of leptomeningeal disease.
Brain Metastases at Diagnosis | Up to 24 Months
  Average number of lesions on diagnostic MRI.
Size of Largest Brain Metastasis | Up to 24 Months
  Average size of largest brain metastasis.
Overall Survival After Brain Metastasis Diagnosis | Up to 48 Months
  Time from brain metastasis diagnosis to death from any cause.
Brain Metastasis Specific Survival | Up to 48 Months
  Time from brain metastasis diagnosis to death attributable to brain metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Baptist Health South Florida, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided